CLINICAL TRIAL: NCT04500769
Title: Muscle-derived Extracellular Vesicles and Their Interactions With Adipocytes in Human Metabolic Dysfunction
Brief Title: Training Induced Muscle Exosome Release
Acronym: TIMER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuan Wen (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Yuan Wen, Assistant Professor, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 43910; 3R01DK119619-02S1 (NIH)
Record Dates: First submitted 2020-07-29; First posted 2020-08-05 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Metabolism
Keywords: Metabolism; Muscle; Extracellular Vesicles; Exosomes; Resistance Exercise
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute Resistance Exercise (Experimental): Participants will perform four exercises: squat, knee extension, leg press, and lat pulldown at 80% of 1-RM determined during a previous visit.
  Interventions: Behavioral: Acute Resistance Exercise

INTERVENTIONS:
Behavioral: Acute Resistance Exercise — Participants will perform three sets of eight repetitions, with a 90-120 second rest between sets, with a fourth set performed to failure. All resistance exercise will be performed on pneumatic resistance devices (Keiser Sports Health Equipment, Fresno, CA).
  Other Names: Strength Training

SUMMARY:
The primary objective of this study is to quantify miR-1 release from muscle in extra-cellular vesicles following an acute resistance exercise bout and potential delivery to subcutaneous adipose tissue in young healthy and obese adults.

DETAILED DESCRIPTION:
Numerous studies in humans and animals have shown that aerobic exercise is beneficial to adipose tissue function and whole-body metabolism. Both acute and chronic aerobic exercise enhance adipocyte catecholamine sensitivity in humans and animals. Although relatively few studies have investigated whether adipose adrenergic signaling is affected by resistance exercise (RE), it is known that a single bout of RE can increase circulating NEFA and resting energy expenditure and decrease respiratory quotient for up to 24 hours, indicative of increased adipocyte lipolysis and muscle fatty acid oxidation. Furthermore, the lipolytic response to RE is impaired in obese men. Using synergist ablation, a model of RE in mice, the investigators show that adipose transcriptional responses are exosome-dependent, and that serum exosomes enhance adipocyte catecholamine sensitivity and lipolysis for at least 24 hours. To the investigator's knowledge, this is the first demonstration of a potential mechanism whereby RE imparts metabolic adaptations in adipose. Since adipose metabolic function is crucial for determining whole-body metabolic outcomes, the ability of RE-induced exosomes to improve adipose metabolism has significant clinical implications.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age.
* Either BMI <25 or >30.
* Relatively sedentary, reporting no participation in regular (>1 day per week) exercise for at least the past 3 months.
* Non-smoker.

Exclusion Criteria:

* BMI between 25 and 30.
* Evidence or signs and symptoms for cardiovascular disease (previous heart attack, arrhythmias, angina, shortness of breath, extreme fatigue, unusual pain in neck, jaw, throat, upper abdomen, or back, swelling in feet, legs, or ankles).
* Evidence or signs and symptoms of metabolic syndrome or disorder (diagnosis of diabetes or insulin resistance, elevated BP, high fasting blood sugar, abnormal cholesterol or triglyceride levels).
* Chronic aspirin or NSAID use (unless it can be safely stopped prior to the biopsies), and any other use of an anticoagulant (e.g., Coumadin) or history of bleeding including history of hypo- or hyper-coagulation disorders.
* Neurological, musculoskeletal, or other disorder that would preclude safe participation in the weight lifting tasks and all performance tests.
* Any other medical condition that would interfere with testing or increase one's risk of complications during exercise, as judged by the study physician.
* Any other condition or events considered exclusionary by the PI and/or physician, such as non-compliance.
* Lidocaine allergy (1% lidocaine is the local anesthetic used during the muscle biopsy procedure).
* Pregnancy.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McCarthy, Ph.D., Principal Investigator — University of Kentucky; Yuan Wen, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were actively recruited from the University of Kentucky campus as well as from the surrounding Lexington community through local advertisement using IRB approved recruitment flyers or newspaper advertisement. Recruitment occurred between March of 2019 and November 2022.
Pre-assignment Details: Consent and baseline assessments were conducted prior to the resistance exercise intervention. Baseline assessments included demographics, medications, personal health and medical history, vitals, and physical activity readiness. Baseline assessment of strength was also conducted for each resistance exercise so that relative intensity could be standardized for each participant. All participants completed the same resistance exercise bout.
Period: Overall Study
Arm/Group | Acute Resistance Exercise
Started | 38
Completed | 33
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: We studied healthy recreationally active males and females between the ages of 18-39.
Arm/Group | Acute Resistance Exercise
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.71 (5.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: miR-1 Abundance
Description: Exosomal, muscle, and adipose miR-1 abundance will be quantified at baseline and following an acute bout of resistance exercise by qPCR.
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Acute Resistance Exercise
Number analyzed (Participants) | 32
percent change
  Percent change in serum EV miR-1 with exercise | 226 (313)
  Percent change in muscle miR-1 with exercise | 110 (82)
  Percent change in adipose miR-1 with exercise | 286 (464)

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: AEs and SAEs were collected according to the standard definitions used by clinicaltrials.gov.
Arm/Group | Acute Resistance Exercise
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 12/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acute Resistance Exercise (N=38)
Light headed from blood draw (Blood and lymphatic system disorders) | 2 (2)
Nausea during exercise (Nervous system disorders) | 4 (4)
Persistent numbness around biopsy site (Musculoskeletal and connective tissue disorders) | 2 (2)
Blister from steri-strip (Skin and subcutaneous tissue disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT04500769/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT04500769/ICF_000.pdf